CLINICAL TRIAL: NCT03480373
Title: Electronic Cigarette Use During Pregnancy
Status: Completed | Type: Observational
Sponsor: UConn Health (Other)
Collaborators: University of Colorado, Denver (Other); Hartford Hospital (Other); Roswell Park Cancer Institute (Other); Denver Health Medical Center (Other); Baystate Medical Center (Other); East Tennessee State University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Erin Mead-Morse, Assistant Professor, UConn Health
Other Study IDs: 17-180-6; 5R01CA207491-04 (NIH)
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cigarette Smoking-Related Carcinoma
Keywords: Nicotine; Nicotine addiction; Tobacco Use Disorder; Pregnancy; Electronic cigarettes; Cigarettes; Vaping; Carcinoma; Pregnant; Birth Outcomes; E-liquid
MeSH Terms: conditions — Tobacco Use Disorder; Vaping; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim 1: To compare the overall toxicant exposure in pregnant women who use electronic cigarettes (e-cigs, vapor, e-liquid, e-juice, vape, vaping devices) compared to women who smoke conventional cigarettes.

Aim 2. To compare toxicant exposure and birth outcomes among infants born to pregnant women who use e-cigs compared to women who smoke conventional cigarettes.

Aim 3. To explore potential mechanisms by which e-cigs could influence birth weight.

DETAILED DESCRIPTION:
In addition to examining characteristics of pregnant e-cig users as well as patterns of their product use, this study is innovative in several ways. First, it is the first known study to examine toxicant exposure to cigarettes and e-cigs in a sample of pregnant smokers who are using these products. Although studies have reported on toxic exposures with e-cigs, this is the first study to apply toxic exposure tests to pregnant women.

Second this is the first study to examine the impact of electronic cigarette use on birth outcomes in pregnant smokers. Although e-cigarettes are similar to tobacco cigarettes in that they deliver nicotine, they are distinguished from tobacco cigarettes in that they do not contain many toxic substances such as carbon monoxide and volatile organic compounds. Consequently, similar to nicotine replacement therapies they have the potential to improve birth outcomes. However, it possible that there may be unanticipated negative effects on birth outcomes, and this study could provide a signal for potential other adverse effects (i.e., miscarriages etc.). Third, this study is the first to examine whether e-cigs alter carcinogen exposure to the fetus, which has been implicated in causing low birth weight and in long-term cancer risk for infants born to smokers. Finally, this is the first study to explore formaldehyde in urine as a measurement of conventional smoking and electronic cigarette use.

ELIGIBILITY:
Inclusion Criteria:

1. cigarette smokers who exclusively smoke conventional cigarettes daily, or who use e-cigs daily, or who use either product daily and the other product at least weekly.
2. Participant is ≤ 24 weeks gestation for conventional smokers and ≤ 36 weeks gestation for e-cig users or dual users.
3. at least 16 years of age
4. able to speak English or Spanish;
5. able to read and sign consent form
6. intent to carry pregnancy to term.

Exclusion Criteria:

1. current drug or alcohol abuse or dependence (other than methadone or buprenorphine maintenance)
2. participant uses combustible marijuana more than 3 times per week (use of edibles/oils is permitted
3. unstable psychiatric disorder
4. unstable medical problems (e.g., pre-eclampsia, threatened abortion, hyperemesis gravidarum)
5. known congenital abnormality
6. Regular use of tobacco products other than conventional or e-cigs

Ages: 16 Years to 45 Years | Sex: Female
Age Groups: Child, Adult
Study Population: * Age: at least 16 years of age
  * Ethnicity: Hispanic and non-Hispanic. All race and ethnic groups will be eligible
  * Gender: Female
  * Other characteristics - (e.g. primary language etc.): English or Spanish speaking
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
To compare the overall toxicant exposure in pregnant women who use electronic cigarettes compared to women who smoke conventional cigarettes. | 9 months
  The overall toxicant exposure will be measured at each trimester and adjusted for potential confounding covariates. A multivariate analysis of variance (MANOVA) with repeated measures will be used to evaluate the pregnant women who use electronic cigarettes compared to women who smoke conventional cigarettes at each trimester.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Mead-Morse, MD, MPH, Principal Investigator — UConn Health
Locations (6):
- United States (6):
  - University of Colorado, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - UCONN Health, Farmington, Connecticut
  - Women's Ambulatory Health Services at Hartford Hospital, Hartford, Connecticut
  - Baystate Medical Center, Springfield, Massachusetts
  - East Tennessee State University, Johnson City, Tennessee